CLINICAL TRIAL: NCT02520466
Title: Effect of Cocoa Flavanol-containing Drink on Coronary Vascular Function in Patients With Coronary Artery Disease
Brief Title: Cocoa Flavanol and Coronary Vasomotion Vascular Function in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EK2012-0201
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Stable Coronary Heart Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- flavanol-containing drink (Active Comparator): flavanol-containing drink
  Interventions: Dietary Supplement: flavanol-rich drink vs flavanol-free drink
- flavanol-free drink (Placebo Comparator): flavanol-free drink matched for taste and calories
  Interventions: Dietary Supplement: flavanol-rich drink vs flavanol-free drink

INTERVENTIONS:
Dietary Supplement: flavanol-rich drink vs flavanol-free drink — Patients will be randomized to either a flavanol-rich drink or a flavanol-free drink of similar volume, taste and calory and sugar content

SUMMARY:
The aim of the present study is to investigate whether the ingestion of a cocoa flavanol-containing drink compared to a flavanol-free drink, improves coronary vasomotion and platelet function in patients with overt coronary artery disease acutely (after 2 hours)

ELIGIBILITY:
Inclusion Criteria:

Patients with coronary artery disease undergoing elective coronary angiography with or without the need of coronary intervention

* Age 20 - 80
* Written obtained informed consent

Exclusion Criteria:

* Acute ST-elevation myocardial infarction
* Acute non-ST-elevation myocardial infarction (enzyme positive)
* Ventricular tachy-arrythmias or AV-Block >I°
* Renal insufficiency (GFR MDRD < 30ml/min) or liver disease (ALT or AST >150 IU)
* Pregnancy
* Known allergy to compounds of cocoa product
* Known allergy to contrast media
* Known allergy to nuts
* Intolerance to coffein and theobromin
* Acute infectious disease
* Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
* Participation in another study within the last month
* Concomitant vitamin supplements and herbal remedies, as well as fruit and tea extracts
* No study visits ± 1 week before Eastern, Christmas and New Year holyday (altered eating habits)
* Extreme eating habits (as assessed by a questionnaire)
* Alcohol or drug abuse
* Lactose intolerance

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
coronary endothelial function as assessed as response to cold pressor test | 2 hours
  Primary endpoint will be the improvement in coronary endothelial function in response to cold pressor testing (i.e. % reduction in coronary artery constriction compared to baseline) 2h after ingestion of a cocoa flavanol rich-drink or placebo drink, respectively.
  In a subset of patients daily consumption of a flavanol-drink will be assessed and outcomes measured after 3-4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Lüscher, Prof MD, Principal Investigator — University Hospital Zurich, Cardiovascular Center Cardiology
Locations (2):
- Switzerland (2):
  - Cardiovascular Center Cardiology Univeristy Hospital of Zurich, Zurich
  - Universisty Hospital of Zurich, Cardiovascular Center Cardiology, Zurich